CLINICAL TRIAL: NCT03457636
Title: The Use of Oracea and Epiduo Forte in Severe Acne Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derm Research, PLLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORA-1801
Record Dates: First submitted 2018-02-27; First posted 2018-03-07 (Actual); Results first posted 2019-03-20 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Doxycycline; Adapalene; Adapalene, Benzoyl Peroxide Drug Combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- doxycycline anhydrous and adapalene/benzoyl peroxide (Experimental): All subjects will receive at Baseline doxycycline anhydrous 40 mg (Oracea) to be taken once daily and Adapalene-Benzoyl Peroxide Gel .3-2.5% (Epiduo) to be applied once daily for 12 weeks
  Interventions: Drug: Doxycycline Anhydrous 40 MG; Drug: Adapalene/Benzoyl Peroxide Gel 0.3-2.5%

INTERVENTIONS:
Drug: Doxycycline Anhydrous 40 MG — One Oracea Capsule (40 mg) should be taken once daily in the morning on an empty stomach, preferably at least one hour prior to or two hours after meals
  Other Names: Oracea
Drug: Adapalene/Benzoyl Peroxide Gel 0.3-2.5% — Epiduo Forte should be applied in a thin layer to affected areas of the face and/or trunk once daily after washing, with care taken to avoid the eyes, lips, and mucous membranes
  Other Names: Epiduo Forte 0.3%-2.5% Topical Gel

SUMMARY:
This is a single-center, open label pilot study. The study is comprised of 5 study visits; Screening, Baseline, and weeks 4, 8, and 12. All subjects will receive Oracea once daily (QD) and Epiduo Forte at Baseline. We will evaluate Investigator Global Assessment (IGA), total lesion count, inflammatory lesion count, non-inflammatory lesion count, adverse events and concomitant medications.

DETAILED DESCRIPTION:
This is a single-center, open label pilot study. The study is comprised of 5 study visits; Screening, Baseline, and weeks 4,8, and 12. All subjects will receive Oracea once daily (QD) and Epiduo Forte at Baseline. WE will evaluate Investigator Global Assessment (IGA), total lesion count, adverse events and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

i. Outpatient, male or female subjects of any race, and at least 12 years of age or older. Female subjects of childbearing potential must have a negative urine pregnancy test result at Baseline (test must have a sensitivity of at least 25 milli-international units/milliliter [mIU/ml] for human chorionic gonadotropin) and practice a reliable method of contraception throughout the study:

A female is considered of childbearing potential unless she is:

* postmenopausal for at least 12 months prior to study drug administration;
* without a uterus and/or both ovaries; or
* has been surgically sterile for at least 6 months prior to study drug administration

Reliable methods of contraception are:

* hormonal methods or intrauterine device in use ≥90 days prior to study drug administration;
* barrier methods plus spermicide in use at least 14 days prior to study drug administration; or
* vasectomized partner (vasectomy must be performed 3 months prior to first study drug administration or in the alternative a zero sperm count will suffice) [Exception: female subjects of childbearing potential who are not sexually active will not be required to practice a reliable method of contraception. These subjects may be enrolled at the Investigator's discretion if they are counseled to remain sexually inactive during the study and understand the possible risks in getting pregnant during the study.] ii. Facial acne IGA score of 4 iii. Minimum of 20 or more inflammatory lesions and 20 or more non-inflammatory lesions and not more than 4 nodules iv. Able to understand the requirements of the study and sign Informed Consent/HIPAA Authorization forms. Subjects under the legal age of consent in the state where the study is conducted must also have the written, informed consent of a parent or legal guardian

Exclusion Criteria:

i. Female subjects who are pregnant (positive urine pregnancy test ), breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control ii. Allergy or sensitivity to any component of the test medication iii. Subjects who have not complied with the proper wash-out periods for prohibited medications (Supplement I)> iv. Medical condition that, in the opinion of the investigator, contraindicates the subject's participation in the clinical study v. Skin disease/disorder that might interfere with the diagnosis or evaluation of acne vulgaris vi. Evidence of recent alcohol or drug abuse vii. History of poor cooperation, non-compliance with medical treatment, or unreliability viii. Exposure to an investigational drug study within 30 days of the Baseline Visit -

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon H. Kircik, M.D., Principal Investigator — Skin Sciences, PLLC
Locations (1):
- Skin Sciences, PLLC, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxycycline Anhydrous 40 mg Once Daily and Adapalene/Benzoyl p: All subjects will receive at Baseline doxycycline anhydrous 40 mg and Adapalene-Benzoyl Peroxide Gel .3-2.5% (Epiduo) to be applied once daily
  Doxycycline Anhydrous 40 MG: One Oracea Capsule (40 mg) should be taken once daily in the morning on an empty stomach, preferably at least one hour prior to or two hours after meals
  Adapalene-Benzoyl Peroxide Gel 0.3-2.5%: Epiduo Forte should be applied in a thin layer to affected areas of the face and/or trunk once daily after washing, with care taken to avoid the eyes, lips, and mucous membranes
Period: Overall Study
Arm/Group | Doxycycline Anhydrous 40 mg Once Daily and Adapalene/Benzoyl p
Started | 22
Completed | 20
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Doxycycline Anhydrous and Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 19 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment (IGA) Score
Description: The IGA is an assessment by the Investigator to assess the severity of the subject's disease wherein 0=Clear Skin, 1=Almost Clear, 2=Mild Severity, 3=Moderate, 4=Severe, 5=Very Severe. Lower score indicate less severe disease.
Time Frame: Baseline, Week 4, Week 8, Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Doxycycline Anhydrous and Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 20
Participants
  Baseline: Almost Clear | 0
  Baseline: Clear | 0
  Baseline: Severe | 20
  Baseline: Moderate | 0
  Baseline: Mild | 0
  Week 4: Almost Clear | 0
  Week 4: Clear | 0
  Week 4: Severe | 5
  Week 4: Moderate | 15
  Week 4: Mild | 0
  Week 8: Almost Clear | 2
  Week 8: Clear | 0
  Week 8: Severe | 0
  Week 8: Moderate | 10
  Week 8: Mild | 8
  Week 12: Almost Clear | 6
  Week 12: Clear | 0
  Week 12: Severe | 0
  Week 12: Moderate | 1
  Week 12: Mild | 13

2. Secondary Outcome: IGA Score
Description: The percent of subjects who have at least a 2 grade improvement on IGA score
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Doxycycline Anhydrous and Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 20
Participants | 19

3. Secondary Outcome: Inflammatory Lesion Count
Description: Inflammatory lesions here include papules and pustules on the face from edge of hairline to mandibular line as counted by the Investigator. Lower counts indicate less severe disease.
Time Frame: Baseline, Week 4, Week 8, Week 12
Measure: Median (Standard Deviation); unit: count of lesions
Arm/Group | Doxycycline Anhydrous and Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 20
count of lesions
  Baseline | 33 (7)
  Week 4 | 21 (6)
  Week 8 | 12 (5)
  Week 12 | 6 (4)

4. Secondary Outcome: Non-inflammatory Lesion Count
Description: Non-inflammatory lesions here include open and closed comedones. These are counted on the face by the investigator from edge of hairline to mandibular line and lower count indicates less severe disease.
Time Frame: Baseline, Week 4, Week 8, Week 12
Measure: Median (Standard Deviation); unit: lesion count
Arm/Group | Doxycycline Anhydrous and Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 20
lesion count
  Baseline | 33 (7)
  Week 4 | 27 (7)
  Week 8 | 17 (7)
  Week 12 | 9 (6)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Doxycycline Anhydrous and Adapalene/Benzoyl Peroxide
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline Anhydrous and Adapalene/Benzoyl Peroxide (N=20)
generalized sunburn (Skin and subcutaneous tissue disorders) | 1 (1)
fracture right foot (Musculoskeletal and connective tissue disorders) | 1 (1)
sinus infection (Infections and infestations) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
rash between and under breasts (Skin and subcutaneous tissue disorders) | 1 (1)
sunburn on face (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT03457636/Prot_SAP_000.pdf